CLINICAL TRIAL: NCT04882111
Title: ALIGN - A Palliative Care Social Work Intervention for Cancer Patients Discharging to a Skilled Nursing Facility
Brief Title: ALIGN Intervention in Patients With Advanced Cancer Discharging to a SNF
Acronym: ALIGN
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 20-1656.cc; P30CA046934 (NIH)
Record Dates: First submitted 2020-11-03; First posted 2021-05-11 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Cancer
Keywords: Palliative
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Discharged Cancer Patients (Experimental): 25 patients, adults ≥ 18, with stage II - IV solid tumor malignancy discharging from an acute care hospital to a SNF in the metro Denver area who have decisional capacity to consent and are English speaking.
  Interventions: Behavioral: ALIGN

INTERVENTIONS:
Behavioral: ALIGN — The ALIGN intervention was developed by the Holding Group, an independent partnership of palliative care-trained social workers. The intervention is theory driven, patient/caregiver centered, addresses palliative care and psychosocial issues, and integrates with health care teams. Working in collaboration with KPCO and Dr. Stacy Fischer (primary mentor), the Holding Group tested the ALIGN intervention in the LTAC and SNF setting (Preliminary Studies). The Holding Group will be the intervention personnel providing psychosocial care that targets communication, goal alignment, and caregiver support.

SUMMARY:
This is a single arm, pre-post, pilot study assessing the feasibility and acceptability of the ALIGN intervention in metastatic adult cancer patients discharging to local area SNFs.

DETAILED DESCRIPTION:
A novel approach for delivering high quality palliative care for cancer patients discharging to a skilled nursing facility (SNF) is critically needed. This investigator plans to test a palliative care social work led intervention called ALIGN (Assessing and Listening to Individual Goals and Needs) that aims to define patient and caregiver goals, facilitate communication between patients and their care teams, and develop a patient-centered plan that accompanies the patient across all future health system transitions. The central hypothesis is that implementation of ALIGN is feasible and acceptable for cancer patients and their caregivers and SNF staff.

ELIGIBILITY:
Inclusion Criteria:

1. Stage II - IV solid tumor malignancy
2. Discharging from an acute care hospital to a SNF in the metro Denver area
3. Decisional capacity to consent
4. English speaking
5. (During COVID requirements) Either internet access through a computer, tablet, or smartphone OR cellular service with adequate allowance of cellular minutes to allow virtual visits (by participant's assessment)

Exclusion Criteria:

1. Discharging with hospice as their goal of care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Subject retention | Two Years
  This investigator anticipates the study to be feasible if enrollment and retention rates of patients and caregivers are within 60% of the goal and if, of those enrolled, 70% of patients and caregivers complete the intervention.

SECONDARY OUTCOMES:
Qualitative interviews of ALIGN participants | 1.5 years
  Study staff will conduct individual semi-structured interviews with 15 patients and 15 caregivers who receive the ALIGN intervention.
Qualitative interviews of SNF staff | 1.5 years
  Exit interviews will be conducted with 10 SNF front line staff (social worker, medical director, care manager, director of nursing) from SNF's that had 2 or more patients that received the intervention.

OTHER OUTCOMES:
Advanced Illness Coordinating Care Survey | Baseline and 60 days
  A survey of satisfaction with care for patients and caregivers
Goal alignment measurement | Baseline and 60 days
  Patients and providers will be asked a focus of treatment question ("Please select one of the options below that best describes your current focus of treatment") and asked to select from the following options: curative, life prolonging/rehabilitative, or comfort focused. Patients and providers will be asked this question at the beginning and end of the study. We are measuring whether there is increased congruence in the response between patient and providers at the end of the study. If there is increased congruence this suggests that the ALIGN intervention is helping facilitate illness and prognostic understanding.
FACIT-Pal | Baseline and 60 days
  This 39 item questionnaire measures four primary quality of life domains: physical well-being, social/family well-being, emotional well-being, functional well-being, and spiritual well-being. Lower scores indicate lower quality of life.
Advance Care Planning documentation | Baseline and 60 days
  Study staff will collect patient and caregiver reported outcomes (virtually by phone or Zoom) to help guide future estimations of sample size. MDPOA, CPR directive, MOST are documents that communicate end of life wishes for patients and also who they would designate to make medical decisions on their behalf if they are unable to do so themselves. We are measuring completion rates of these documents in patients who participate in the ALIGN intervention. The more patients that have an MDPOA/CPR directives/MOST form completed after the intervention suggests that the ALIGN intervention helps people with advance care planning.
Decision Regret Scale | Baseline and 60 days
  This 5 item scale measures distress or remorse after a health care decision. The minimum score is 0 and the maximum score is 100. A higher score indicates greater regret.
Caregiver Reaction Assessment | Baseline and 60 days
  This is a 24 item instrument designed to measure the reactions of family members to caring for adults with a variety of illness. The instrument focuses on five dimensions: caregiver's esteem, lack of family support, impact on finances, impact on schedule, and impact on health. The minimum score is 0 and the maximum score is 24. A higher score indicates greater caregiver burden.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Singh S, Dafoe A, Lahoff D, Tropeano L, Owens B, Nielsen E, Cagle J, Lum HD, Dorsey Holliman B, Fischer S. A Process Evaluation of a Palliative Care Social Work Intervention for Cancer Patients in Skilled Nursing Facilities. J Palliat Med. 2024 Jun;27(6):734-741. doi: 10.1089/jpm.2023.0381. Epub 2024 Apr 2. PMID 38563805
- [Derived] Singh S, Dafoe A, Lahoff D, Tropeano L, Owens B, Nielsen E, Cagle J, Lum HD, Dorsey Holliman B, Fischer S. Pilot Trial of a Social Work Intervention to Provide Palliative Care for Adults with Cancer in Skilled Nursing Facilities. J Palliat Med. 2023 Apr;26(4):527-538. doi: 10.1089/jpm.2022.0413. Epub 2022 Nov 21. PMID 36409676